CLINICAL TRIAL: NCT00118638
Title: A Randomized, Double Blind, Active-Controlled Study of Darbepoetin Alfa for the Treatment of Anemia in Subjects With Non-Myeloid Malignancy Receiving Multicycle Chemotherapy
Brief Title: A Study of Darbepoetin Alfa for the Treatment of Anemia in Subjects With Non-Myeloid Malignancy Receiving Multicycle Chemotherapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20030231
Record Dates: First submitted 2005-06-30; First posted 2005-07-12 (Estimated); Last update posted 2013-04-29 (Estimated); Status verified 2013-04

CONDITIONS: Anemia; Non-Myeloid Malignancies
Keywords: Non-myeloid malignancy; Darbepoetin alfa; Clinical Trial
MeSH Terms: conditions — Anemia | interventions — Darbepoetin alfa

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Darbepoetin alfa 500 mcg - Group A (Experimental)
  Interventions: Drug: Darbepoetin alfa - 500mcg
- Darbepoetin alfa 2.25 mcg/kg - Group B (Active Comparator)
  Interventions: Drug: Darbepoetin alfa - 2.25 mcg/kg

INTERVENTIONS:
Drug: Darbepoetin alfa - 2.25 mcg/kg — Darbepoetin alfa 2.25 mcg/kg QW dosing/ placebo Q3W
  Arms: Darbepoetin alfa 2.25 mcg/kg - Group B
Drug: Darbepoetin alfa - 500mcg — Darbepoetin alfa 500mcg Q3W dosing / placebo QW
  Arms: Darbepoetin alfa 500 mcg - Group A

SUMMARY:
The purpose of this study is to evaluate the efficacy of darbepoetin alfa as 500ug once every 3 weeks to show that the dose and schedule are not inferior to darbepoetin alfa administered as 2.25ug/kg once per week in the treatment of anemia in subjects with non-myeloid malignancies.

ELIGIBILITY:
Inclusion Criteria:

* Non-myeloid malignancy
* At least 12 additional weeks of cyclic cytotoxic chemotherapy anticipated regardless of schedule
* Eastern Cooperative Oncology Group performance status of 0-2
* Hemoglobin concentration of less than 11 g/dL within 24 hours before randomization
* Of legal age at the time written informed consent is obtained

Exclusion Criteria:

* Known history of seizure disorder
* Known primary hematologic disorder, which could cause anemia, other than a non-myeloid malignancy
* Unstable or uncontrolled disease/condition, related to or affecting cardiac function
* Clinically significant inflammatory disease
* Inadequate renal and/or liver function
* Known positive HIV test
* Previously suspected of or confirmed to have neutralizing antibodies to rHuEPO
* Received more than 2 red blood cell (RBC) transfusions within 4 weeks before randomization or any RBC transfusion within 14 days before randomization, or any planned RBC transfusion between randomization and study day 1
* Received any erythropoietic therapy within 4 weeks before randomization or any planned erythropoietic therapy between randomization and study day 1
* Other investigational procedures
* Subject is currently enrolled in or less than 30 days since receipt of any investigational drug or device that is not approved by the applicable regulatory authority
* Pregnant or breast feeding
* Not using adequate contraceptive precautions
* Known sensitivity to any of the products to be administered during dosing
* Previously randomized in this study
* Concerns for subject's compliance with protocol procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 705 (Actual)
Dates: Start 2004-03; Primary Completion 2004-12 (Actual); Study Completion 2005-01 (Actual)

PRIMARY OUTCOMES:
Incidence of at least one RBC transfusion from week 5 to End of Treatment Period (EOTP) | from week 5 to EOTP

SECONDARY OUTCOMES:
Incidence of achieving a hemoglobin concentration of greater than or equal to 11.0 g/dL, in the absence of RBC transfusions in the preceding 28 days, from week 5 to EOTP | from week 5 to EOTP
Incidence of at least one RBC transfusion from week 1 (day 1) to EOTP | from week 1 (day 1) to EOTP
Incidence of achieving a hemoglobin concentration greater than or equal to 11.0 g/dL, in the absence of RBC transfusions in the preceding 28 days, from week 1 to EOTP | from week 1 to EOTP
Change in FACT-G Physical Well-being subscale from baseline to EOTP | from baseline to EOTP
Change in hemoglobin from baseline to EOTP | from baseline to EOTP
Change in FACT-Fatigue subscale score from baseline to EOTP | from baseline to EOTP
Change in FACT-G total score from baseline to EOTP | from baseline to EOTP
Change in EQ-5D Thermometer from baseline to EOTP | from baseline to EOTP
Change in BSI Anxiety scale score from baseline to EOTP | from baseline to EOTP
Change in BSI Depression scale score from baseline to EOTP | from baseline to EOTP
Incidence and severity of adverse events | throughout study
Incidence of hemoglobin concentration greater than 13.0 g/dL at any time on study | at any time on study
Change in number of caregiver hours from baseline to EOTP | from baseline to EOTP
Incidence of an increase in hemoglobin concentration greater than or equal to 2 g/dL in a 28-day window and any negative clinical consequences | throughout study
Incidence of an increase in hemoglobin concentration of greater than or equal to 1 g/dL in a 14-day window and any negative clinical consequences | throughout study
Incidence of a confirmed antibody formation to darbepoetin alfa | throughout study

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Background] Canon JL, Vansteenkiste J, Hedenus M, Gascon P, Bokemeyer C, Ludwig H, Vermorken J, Legg J, Pujol B,
- [Result] Canon JL, Vansteenkiste J, Hedenus M, Gascon P, Bokemeyer C, Ludwig H, Vermorken J, Legg J, Pujol B, Bridges K. Transfusion risk in cancer patients with chemotherapy-induced anemia when initiating darbepoetin alfa therapy at a baseline hemoglobin level of <9 g/dL versus 9 to <10 g/dL versus >/= 10 g/dL: an exploratory analysis of a phase 3 trial. Med Oncol. 2012 Sep;29(3):2291-9. doi: 10.1007/s12032-011-0103-x. Epub 2011 Nov 13. PMID 22081263
- [Result] Canon JL, Vansteenkiste J, Bodoky G, Mateos MV, Bastit L, Ferreira I, Rossi G, Amado RG. Randomized, double-blind, active-controlled trial of every-3-week darbepoetin alfa for the treatment of chemotherapy-induced anemia. J Natl Cancer Inst. 2006 Feb 15;98(4):273-84. doi: 10.1093/jnci/djj053. PMID 16478746
- [Result] Vansteenkiste J, Hedenus M, Gascon P, Bokemeyer C, Ludwig H, Vermorken J, Hamilton L, Bridges K, Pujol B. Darbepoetin alfa for treating chemotherapy-induced anemia in patients with a baseline hemoglobin level < 10 g/dL versus > or = 10 g/dL: an exploratory analysis from a randomized, double-blind, active-controlled trial. BMC Cancer. 2009 Sep 3;9:311. doi: 10.1186/1471-2407-9-311. PMID 19728887
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com
- See also: Notice regarding posted summaries of trial results — http://download.veritasmedicine.com/REGFILES/amgen/Amgen_results_disclaimer.pdf
- See also: To access clinical trial results information click on this link — http://download.veritasmedicine.com/REGFILES/amgen/20030231.pdf
- See also: FDA-approved Drug Labeling — http://www.aranesp.com/